CLINICAL TRIAL: NCT04077918
Title: Comparison of the Effects of Animal Protein Diet and Plant Protein Diet on Blood Test Result and Clinical Outcome in Hemodialysis Patients
Brief Title: Comparison of the Effects of Different Protein Diet in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Camillians Saint Mary's Hospital Luodong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SMHprotdiet
Record Dates: First submitted 2019-08-24; First posted 2019-09-04 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diffenence of Protein Diets on Hemodialysis Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant protein diet (Active Comparator): 18 g of plant protein diet added every day for 3 months , and after washout for 1 month, 18 g of animal protein diet added every day for 3 months
  Interventions: Dietary Supplement: protein diet
- Animal protein diet (Active Comparator): 18 g of animal protein diet added every day for 3 months, and after washout for 1 month, 18 g of plant protein diet added every day for 3 months
  Interventions: Dietary Supplement: protein diet

INTERVENTIONS:
Dietary Supplement: protein diet — 100 CHD patients will be recruited and randomized into 2 groups with an additional animal or plant protein 18g per day

SUMMARY:
Chronic hemodialysis (CHD) patients are vulnerable to develop protein energy malnutrition and make a notion that to maintain the nutritional status is of paramount importance in these patients. However, proteins intake from vegetarian and meat diet were observed to have different impacts on nutritional and inflammatory status, mineral homeostasis and its related hormones, and clinical outcomes in non-dialysis CKD patients. In here, we aim to investigate these impacts in CHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patient

Exclusion Criteria:

1. Hemodialysis less than 3 months
2. Age < 20 years or >90 years
3. Serum albumin < 3 g/dL，
4. Daily protein diet < 0.6 gm/kg/day or > 1.2 gm/kg/ day，
5. Cannot obey the diet plan: Gastrectomy, difficult in swallowing
6. Active infection, severe illness: cancer patient, liver cirrhosis, etc.
7. Unable to cooperate in the study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Statistical difference of serum biomarkers ( P value) | 7 months
  The items scheduled to be evaluated in this study include serum albumin, pre-albumin, phosphate, calcium, magnesium, lipid profile, ferritin, transferrin, hs-CRP, Alk-P, iPTH, 25(OH)D3, intact & C-terminal FGF23, Klotho and hepcidin levels. We'll collect the patient's serum data in plant diet group, and collect the serum data in animal diet group, then we'll compare the data in these two groups to see whether there is any difference between each item.

SECONDARY OUTCOMES:
Statistical difference of medical visits | 7 months
  We'll review the patient's medical record in outpatient department . We'll look at what's the diagnosis and what's the number of the medical visits during the study period.

OTHER OUTCOMES:
Statistical difference of admissions | 7 months
  . We will also review the patient's admission record to see what's the diagnosis and what's the number of admission during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ching Tsai, MD, Principal Investigator — St. Mary's Hospital Luodong

IPD SHARING:
Plan to Share IPD: No